CLINICAL TRIAL: NCT07130864
Title: Early Vs Late Laparoscopic Cholecystectomy After Ercp For Choledocholithiasis, A Randomised Control Trial.
Brief Title: Early vs Late Laparoscopic Cholecystectomy After Common Bile Duct Stones Clearance Through Ercp.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr Saeed Sarwar, Doctor, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 530/DME/KMC
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Cholecystectomy; Choledocholithiasis; ERCP; Bile Duct Injury
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Group (Experimental): Early group consist of those patients whose cholecystectomy is performed within 72 hours of ERCP .
  Interventions: Procedure: Early cholecystectomy
- Late group (Experimental): Late group consist of those patients whose cholecystectomy is performed after 72 hours of ERCP.
  Interventions: Procedure: Late cholecystectomy

INTERVENTIONS:
Procedure: Early cholecystectomy — Early cholecystectomy is performed within 72 hours of ERCP.
  Arms: Early Group
Procedure: Late cholecystectomy — Late cholecystectomy is performed after 72 hours of ERCP
  Arms: Late group

SUMMARY:
There is controversy about timing of cholecystectomy after the common bile duct is cleared of stones. our study aims to compare the results of early vs late cholecystectomy.

ELIGIBILITY:
Inclusion criteria :

.All patients undergoing laparoscopic cholecystectomy who had concomitant choledocholithiasis for which ercp is done.

exclusion criteria:

.Non consenting indviduals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difficulty level of cholecystectomy | From start of surgery till end, On day 1 of surgery
  the presence of diffuse pericholecystic scar adhesions, Calot's triangle with intense fibrosis, atrophic gallbladder, presence of a cholecysto-enteric or cholecyto-choledochal fistula, presence of necrotic changes, liver abscess or the presence of impacted stones and the help of a senior colleague will be considered a difficult cholecystectomy

SECONDARY OUTCOMES:
Bile duct injury | From the day 1 of surgery till one month
  Bile duct injury that ocuurs intraoperatively or detected in postoperative period
Hospital stay | from day 1 of surgery till discharge, upto 1 month
  Hospital stay determined from day of surgery till discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber teaching hospital, Peshawar, Khyberpukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patients confidentiality maybe breached